CLINICAL TRIAL: NCT03779828
Title: A Multicenter Pilot Study to Determine Criteria for Evaluating the Effectiveness of Two Comparative Monitoring Methods in the Management of Patients With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Receiving Home-based Treatment With IVIg (Privigen®)
Brief Title: Evaluating the Effectiveness of Telemonitoring System in the Management of Patients With CIDP
Acronym: HELIPAD 1
Status: Terminated | Type: Observational
Why Stopped: Due to logistical concerns
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: IgPro10_5004; 2016-A00147-44 (Other: ANSM)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: CIDP; Telemonitoring; Telemedicine
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HOME LINK — Telemonitoring system which include web platform and connected devices.

SUMMARY:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a chronic demyelinating polyneuropathy of autoimmune origin with a progressive or relapsing course.

Diagnosis is based on clinical presentation and electrophysiological findings in accordance with the EFNS/PNS consensus guidelines. IVIg is the first line treatment witch has been shown to be effective in several placebo-controlled trials.

Once IVIg therapy produces a response and is well tolerated, some patients are able to continue their treatment in the home setting. The HOME LINK system offers an integrated, global solution based on telemonitoring technology providing continuous, remote monitoring of Privigen® infusions administered at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of CIDP as per EFNS/PNS criteria.
* Patient already receiving home-based treatment with Privigen®

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving home-based IVIg therapy with Privigen
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Evaluate HOME LINK telemonitoring system for patients receiving home-based IVIg therapy | 52 weeks
  The conventional method of home monitoring requires using a visiting nurse. HOME LINK is a telemonitoring system that is an alternative to this conventional method offering remote at-home monitoring. HOME LINK monitors the patient's health parameters from home. In this way it enables an adjustment of the infusion conditions or intervention of a qualified healthcare professional in the event of an incident. Home Link will be evaluated for failure rate of connection to the telemonitoring platform, failure rate of transmission of self-measurements to the telemonitoring platform, failure rate of transmission of documents relating to home-based treatment, and failure rate of contacting one of the healthcare professionals involved in patient care during the at-home infusions.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Hôpital Pellegrin, Bordeaux University Hospital (CHU), Bordeaux
  - Hôpital Henri Mondor - APHP, Créteil
  - Hôpital Roger Salengro - CHRU, Lille
  - Hôpital Pierre Wertheimer - HCL, Lyon
  - Hôpital La Timone - APHM, Marseille
  - Hôpital Gui de Chauliac - Montpellier University Hospital (CHU), Montpellier
  - Hôpital Pasteur 2 - Nice University Hospital (CHU), Nice
  - Hôpital La Pitié-Salpêtrière - APHP, Paris
  - Hôpital Lariboisière - APHP, Paris
  - Hôpital Nord - Saint Etienne University Hospital (CHU), Saint-Etienne

IPD SHARING:
Plan to Share IPD: No